CLINICAL TRIAL: NCT07008339
Title: Impact of Nipple Reconstruction in Mastectomized Patients Using Cross-Linked Hyaluronic Acid Injection.
Acronym: RECHIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-23-109
Record Dates: First submitted 2025-05-22; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms; Mastectomy; Mammaplasty; Nipple Disorder; Tattooing; Hyaluronic Acid; Dermal Fillers; Reconstructive Surgical Procedures; Quality of Life; Self Concept; Body Image; Patient Satisfaction; Breast Reconstruction; Nipple Reconstruction
Keywords: Breast Cancer; Mastectomy; Breast Reconstruction; Nipple-Areola Complex Reconstruction; Nipple Reconstruction; Areola Reconstruction; Hyaluronic Acid; Dermal Fillers; Micropigmentation; Tattooing; Body Image; Quality of Life; Postmastectomy Reconstruction; Cross-linked Hyaluronic Acid; Patient Satisfaction; Breast Cancer Survivors
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Mixed-methods study with a sequential explanatory design. Phase 1: Quantitative methodology. A parallel, randomized clinical trial developed based on the following hypothesis: nipple reconstruction using hyaluronic acid injection and micropigmentation increases satisfaction and quality of life in mastectomized patients.
  Phase 2: Qualitative methodology. Constructivist paradigm. Descriptive phenomenological study.
  The study will be conducted at the Areolar Micropigmentation Unit (UMA) of Germans Trias i Pujol University Hospital, a high-technology public hospital in the province of Barcelona, serving a local population of 250,000 and acting as a referral center for over 800,000 people. The UMA, part of the Breast Pathology Service and collaborating with the Plastic Surgery Department, treats an average of 53 patients per year and is staffed by two nurses specialized in Body Image and Dermoaesthetics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micropigmentation Only (Active Comparator): Participants receive only areola micropigmentation.
  Interventions: Procedure: Areola Micropigmentation
- Micropigmentation Plus Hyaluronic Acid Filler (Experimental): Participants receive areola micropigmentation and hyaluronic acid filler injection to restore nipple projection.
  Interventions: Device: Hyaluronic Acid Filler Injection

INTERVENTIONS:
Procedure: Areola Micropigmentation — Areola micropigmentation performed by trained nurses
  Arms: Micropigmentation Only
Device: Hyaluronic Acid Filler Injection — Subcutaneous injection of cross-linked hyaluronic acid filler (Juvederm®) for nipple projection.
  Arms: Micropigmentation Plus Hyaluronic Acid Filler

SUMMARY:
This study evaluates the impact of hyaluronic acid (HA) injection for nipple projection following mastectomy, as a complement to areola micropigmentation. While micropigmentation is standard in nipple-areola complex (NAC) reconstruction, HA use remains novel, with limited data on psychosocial, sexual, and aesthetic outcomes.

A sequential explanatory mixed-methods design will be used. In Phase 1, a randomized controlled trial will compare two groups: one receiving NAC micropigmentation alone (control) and the other receiving micropigmentation plus HA-based nipple projection (intervention). A total of 138 participants will be recruited at the Areolar Micropigmentation Unit of Germans Trias i Pujol University Hospital (Barcelona) over 36 months. Outcomes will include psychosocial and sexual well-being, satisfaction with breast and nipple appearance, and nipple projection, measured using the Spanish BREAST-Q, a custom satisfaction tool, and calipers.

Phase 2 will involve a qualitative phenomenological study using semi-structured interviews with a purposive sample from the intervention group. Thematic analysis will explore body image, emotional and social well-being, and overall satisfaction, using NVivo software.

This is the first study assessing HA nipple reconstruction by advanced practice nurses using validated patient-reported outcomes. While the BREAST-Q is appropriate, it may not fully capture emotional nuances, justifying qualitative exploration. HA durability is estimated at 6-9 months, but residual volume and satisfaction over time remain underexplored. HA's aesthetic footprint may allow reduced dosages in future applications.

This minimally invasive technique may reduce the need for surgical nipple reconstruction. Conducting the procedure in a nurse-led setting is novel and may enhance patient-centered care and the role of nursing in post-mastectomy recovery.

The study complies with the Declaration of Helsinki and Spanish biomedical regulations. Ethical approval was obtained. Participants will provide informed consent, and data will be anonymized and securely stored.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant neoplasm among women worldwide. Similarly, in Spain, it is also the most prevalent tumor in women, surpassing colorectal cancer. The incidence of this disease in our country has steadily increased over the past decades, with approximately 26,000 cases diagnosed each year, accounting for 25-30% of all female malignancies. For affected individuals, both the disease and its treatment lead to physical and bodily changes, which in turn have significant emotional implications. A woman facing a breast cancer diagnosis and its associated management goes through a critical period in her life. During this time, the altered self-image resulting from various treatment side effects is often accompanied by a fear of losing femininity and self-confidence, with potentially significant repercussions on the patient's quality of life.

Modern society increasingly demands not only the cure of diseases but also the consideration of factors that enhance patients' quality of life. According to data from the Spanish Society of Plastic, Reconstructive and Aesthetic Surgery (SECPRE), of the 36,000 women mentioned above, approximately 64% will require a mastectomy-defined as the surgical removal of the entire affected breast-and 28% will undergo breast reconstruction.

For these women, the final stage of breast reconstruction typically culminates in the reconstruction of the nipple-areola complex (NAC), which, according to DiCenso et al., represents the conclusion of surgical and adjuvant treatments, as well as the end of uncertainty. It symbolizes the transition from patient to survivor. The healing process is not considered complete until the areola and nipple are reconstructed, thus achieving a morphologically complete breast rather than merely restoring volume.

Micropigmentation is a technique involving the deposition of pigment into the skin using ultra-fine needles. It is simple, safe, does not require general anesthesia, and can be performed by trained nurses in outpatient settings. When a neo-nipple has not been created or has retracted, subcutaneous injection of cross-linked hyaluronic acid (HA) can restore lost volume, improve the realism of micropigmentation, and support emotional healing by improving body image and self-esteem. HA is safe, hydrophilic, biocompatible, and widely used in dermal fillers for volume projection.

This study aims to evaluate the impact of HA-based nipple reconstruction in terms of psychosocial and sexual well-being, satisfaction with the breasts and nipples, and the patient's lived experience.

Specific objectives include:

Identifying the sociodemographic and clinical characteristics of the participants.

Assessing differences in psychosocial and sexual well-being, satisfaction with breasts, nipples, and micropigmentation.

Determining nipple projection and HA retention.

Exploring patient experiences with quality of life, self-confidence, and emotional recovery.

Study Design:

This is a mixed-methods study employing a sequential explanatory design. Phase 1 is a randomized controlled trial comparing micropigmentation alone (control) with micropigmentation plus HA injection (intervention). Phase 2 is a descriptive phenomenological study using semi-structured interviews and thematic analysis.

Setting:

Conducted at the Areolar Micropigmentation Unit, Germans Trias i Pujol University Hospital in Barcelona, a high-tech center that treats 53 patients yearly and is staffed by nurses trained in body image and dermoesthetics.

Population:

Women ≥18 undergoing NAC micropigmentation for the first time. Exclusion criteria include HA allergy or intolerance. Sample size: 138 women (69 per group) in Phase 1. Phase 2 will continue until data saturation (typically 5-15 participants).

Measurements:

BREAST-Q (Spanish version) will assess well-being and satisfaction. A custom questionnaire will assess satisfaction with micropigmentation. Nipple projection will be measured with calipers, and HA data recorded. Interviews will explore body image, self-esteem, intimacy, and expectations.

Data Collection:

Patients will be enrolled during UMA visits. After consent, baseline data and BREAST-Q will be collected. Micropigmentation will be done in 2-4 sessions. For the intervention group, HA will be administered 15 days post-micropigmentation in 2-3 dermal injections. Follow-ups include questionnaires post-procedure and at 3 and 6 months.

Analysis:

Quantitative data will be analyzed using SPSS v.29 with descriptive and inferential statistics (t-test, ANOVA, Mann-Whitney U, chi-square). Qualitative data will be analyzed using Braun & Clarke's method in NVivo. Trustworthiness will be ensured by Lincoln & Guba's criteria.

Limitations:

Challenges include lack of double-blinding, variable timelines, and emotional vulnerability. Measures include standardized protocols and extended data collection.

Justification:

This is the first study to evaluate HA-based nipple reconstruction performed by advanced practice nurses using validated PROMs. HA offers a minimally invasive, adjustable alternative to surgery with fewer complications. Its application in nurse-led outpatient care is novel.

Ethics:

Approved by the Ethics Committee of Germans Trias i Pujol Hospital. Conducted in compliance with the Declaration of Helsinki, Spanish biomedical regulations, and data protection laws (LOPD 3/2018). Informed consent will be obtained. Data will be pseudonymized and securely stored.

ELIGIBILITY:
* Quantitative Phase
* Inclusion Criteria:

Women over 18 years of age, or with parental or legal guardian consent.

At least one of the following criteria:

Women undergoing their first nipple-areola complex (NAC) reconstruction through micropigmentation and/or:

No previous neo-nipple surgery, either unilaterally or bilaterally.

Surgical reconstruction of the areola.

Surgical reconstruction of the NAC with subsequent retraction of the neo-nipple.

More than 6 months since their last surgery.

- Exclusion Criteria:

Allergy to hyaluronic acid.

Poor tolerance to needle injections.

Withdrawal Criteria:

Participant's voluntary decision.

Complications associated with the technique (allergy, hematoma, etc.).

Clinical deterioration preventing the woman from continuing in the study.

- Qualitative Phase

Participant Profile Characteristics: For the qualitative phase, women who have received NAC reconstruction with HA will be invited to participate, following the maximum variation criterion. To ensure the inclusion of participants with diverse characteristics and capture a wide range of perspectives and experiences on the phenomenon under study, women of varying ages, with different breast cancer diagnoses, and histories of various oncological, surgical, and therapeutic treatments will be selected.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2029-07-02 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Nipple Reconstruction | 3, and 6 months after final injection session
  Patient-reported satisfaction with nipple reconstruction, measured using the "Satisfaction with Nipple" scale of the Spanish version of the BREAST-Q questionnaire. This scale ranges from 0 to 100, with higher scores indicating greater satisfaction."

SECONDARY OUTCOMES:
Psychosocial Well-being | Baseline, 3 months, and 6 months post-intervention
  Psychosocial well-being assessed using the 'Psychosocial Well-being' domain of the Spanish version of the BREAST-Q questionnaire. This scale ranges from 0 (lowest well-being) to 100 (highest well-being), with higher scores indicating better psychosocial outcomes.
Sexual Well-being | Baseline, 3 months, and 6 months post-intervention
  Sexual well-being assessed using the 'Sexual Well-being' domain of the Spanish version of the BREAST-Q questionnaire. This scale ranges from 0 (lowest sexual well-being) to 100 (highest sexual well-being), with higher scores indicating better outcomes.
Satisfaction with Breasts | Baseline, 3 months, and 6 months post-intervention
  Satisfaction with breast appearance, measured using the 'Satisfaction with Breasts' subscale of the Spanish version of the BREAST-Q questionnaire. This scale ranges from 0 (lowest satisfaction) to 100 (highest satisfaction), with higher scores indicating better outcomes.
Satisfaction with Micropigmentation | Periprocedural
  Patient-reported satisfaction with areola micropigmentation, measured using a custom satisfaction questionnaire. Higher scores indicate better satisfaction outcomes.
Nipple Projection | Immediately post-procedure, 3 months, and 6 months
  Nipple projection (in mm) measured using digital caliper.
Retention of Hyaluronic Acid | 3 and 6 months post-injection
  Estimated percentage of projection retained over time compared to immediate post-injection measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Huertas Zurriaga, RN, Study Director — Germans Trias i Pujol Hospital; Sergio Alonso Fernández, RN, Study Director — University of Barcelona; Joan Blanco Blanco, RN, Study Director — Universitat de Lleida; Isabel Granados Navarrete, RN, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this trial will be made available, including text, tables, figures, and appendices. Data will be shared beginning 6 months following publication and will be available to researchers who provide a methodologically sound proposal, subject to approval by the study sponsor and ethics committee. Data access will be granted for the purpose of academic research. Proposals should be submitted to [contact email or data request URL].
Supporting Information: Study Protocol, SAP
Time Frame: 6, 12 months after study completion
Access Criteria: Available upon reasonable request and subject to institutional review

REFERENCES:
- [Background] Spear SL, Arias J. Long-term experience with nipple-areola tattooing. Ann Plast Surg. 1995 Sep;35(3):232-6. doi: 10.1097/00000637-199509000-00002. PMID 7503514
- [Background] Halvorson EG, Cormican M, West ME, Myers V. Three-dimensional nipple-areola tattooing: a new technique with superior results. Plast Reconstr Surg. 2014 May;133(5):1073-1075. doi: 10.1097/PRS.0000000000000144. PMID 24776543
- [Background] Martinez P, Jimeno J, Hernanz F, Munoz P. Spanish version of the BREAST-Q(R) 2.0 questionnaire-breast reduction module-: Linguistic, cross-cultural adaptation and validation. Cir Esp (Engl Ed). 2023 Mar;101(3):232-234. doi: 10.1016/j.cireng.2022.10.016. Epub 2022 Oct 18. No abstract available. PMID 36265774
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Moser A, Korstjens I. Series: Practical guidance to qualitative research. Part 3: Sampling, data collection and analysis. Eur J Gen Pract. 2018 Dec;24(1):9-18. doi: 10.1080/13814788.2017.1375091. Epub 2017 Dec 4. PMID 29199486
- [Background] Smallman A, Crittenden T, MiinYip J, Dean NR. Does nipple-areolar tattooing matter in breast reconstruction? A cohort study using the BREAST-Q. JPRAS Open. 2018 Feb 27;16:61-68. doi: 10.1016/j.jpra.2018.01.003. eCollection 2018 Jun. PMID 32158811
- [Background] Beasley KL, Weiss MA, Weiss RA. Hyaluronic acid fillers: a comprehensive review. Facial Plast Surg. 2009 May;25(2):86-94. doi: 10.1055/s-0029-1220647. Epub 2009 May 4. PMID 19415575
- [Background] Kyriazidis I, Spyropoulou GA, Zambacos G, Tagka A, Rakhorst HA, Gasteratos K, Berner JE, Mandrekas A. Adverse Events Associated with Hyaluronic Acid Filler Injection for Non-surgical Facial Aesthetics: A Systematic Review of High Level of Evidence Studies. Aesthetic Plast Surg. 2024 Feb;48(4):719-741. doi: 10.1007/s00266-023-03465-1. Epub 2023 Aug 10. PMID 37563436
- [Background] Ho D, Jagdeo J. Safety and Efficacy of a Volumizing Hyaluronic Acid Filler for Treatment of HIV-Associated Facial Lipoatrophy. JAMA Dermatol. 2017 Jan 1;153(1):61-65. doi: 10.1001/jamadermatol.2016.3827. PMID 27806168
- [Background] Sisti A, Grimaldi L, Tassinari J, Cuomo R, Fortezza L, Bocchiotti MA, Roviello F, D'Aniello C, Nisi G. Nipple-areola complex reconstruction techniques: A literature review. Eur J Surg Oncol. 2016 Apr;42(4):441-65. doi: 10.1016/j.ejso.2016.01.003. Epub 2016 Jan 30. PMID 26868167
- [Background] Boccola MA, Savage J, Rozen WM, Ashton MW, Milner C, Rahdon R, Whitaker IS. Surgical correction and reconstruction of the nipple-areola complex: current review of techniques. J Reconstr Microsurg. 2010 Nov;26(9):589-600. doi: 10.1055/s-0030-1263290. Epub 2010 Aug 18. PMID 20721849
- [Background] Bellman B, von Grote E, Nogueira A. Hyaluronic acid gel filler for nipple enhancement following breast reconstruction. Cutis. 2017 Aug;100(2):107-109. PMID 28961285
- [Background] Panettiere P, Marchetti L, Accorsi D. Filler injection enhances the projection of the reconstructed nipple: an original easy technique. Aesthetic Plast Surg. 2005 Jul-Aug;29(4):287-94. doi: 10.1007/s00266-004-0145-y. PMID 16044237
- [Background] Sue GR, Seither JG, Nguyen DH. Use of hyaluronic acid filler for enhancement of nipple projection following breast reconstruction: An easy and effective technique. JPRAS Open. 2019 Nov 5;23:19-25. doi: 10.1016/j.jpra.2019.10.003. eCollection 2020 Mar. PMID 32158901
- [Background] Ruffolo AM, Bruce WJ, Daugherty THF, Lee J, Sommer NZ. Technical Refinement in Three-Dimensional Nipple-Areola Complex Tattooing of the Reconstructed Breast. Plast Reconstr Surg. 2021 Oct 1;148(4):737-746. doi: 10.1097/PRS.0000000000008390. PMID 34550927
- [Background] DiCenso D, Fischer-Cartlidge E. Nipple-Areola Tattoos: Making the Right Referral. Oncol Nurs Forum. 2015 Nov;42(6):E376-81. doi: 10.1188/15.ONF.E376-E381. PMID 26488844
- [Background] Sehati Shafaee F, Mirghafourvand M, Harischi S, Esfahani A, Amirzehni J. Self-Confidence and Quality of Life in Women Undergoing Treatment for Breast Cancer. Asian Pac J Cancer Prev. 2018 Mar 27;19(3):733-740. doi: 10.22034/APJCP.2018.19.3.733. PMID 29582628